CLINICAL TRIAL: NCT03156946
Title: Breastfeeding Peer Counselling for Mothers of Preterm Neonates: a Stepped- Wedge Cluster Randomized Controlled Trial
Brief Title: Evaluation of a Peer Counseling Breastfeeding Support Program for Mother-preterm Infant Dyads
Acronym: ALAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL17_0033
Record Dates: First submitted 2017-05-02; First posted 2017-05-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Infant Premature
Keywords: breastfeeding; mother-to-mother support; lactation consultant; stepped wedge cluster randomized trial; peer counseling
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Intervention Model Description: stepped wedge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding support program (Experimental)
  Interventions: Behavioral: breastfeeding mother-to-mother support
- Usual or routine care (Other)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: breastfeeding mother-to-mother support — The mother-infant dyads in the intervention arm will receive breastfeeding mother-to-mother support from the hospitalization in the maternity and NICU up to 1 month after discharge. The intervention will be in addition to the usual or routine care. Breastfeeding counselors will be voluntary mothers who breastfed their own preterm infant (aged between 6 months and 5 years at the time of the study) for a minimum of 2 months, and who have had a positive personal breastfeeding experience, and who have undertaken a training course.
  Arms: Breastfeeding support program
Behavioral: Control — The mother-infant dyads in the control arm will continue to receive the usual/routine care provided by participating centers during the hospitalization and Mother and Infant Protection service after discharge.
  Arms: Usual or routine care

SUMMARY:
Breastfeeding has a fundamental impact on the short-, medium- and long-term health of children and has an important impact on women's health. Breastfeeding protects against gastrointestinal and respiratory illnesses and is associated with better cognitive development in childhood, particularly in preterm infants. Despite these potential benefits, preterm infants experience lower rates of breastfeeding initiation and continuation compared to term infants.

The use of breastfeeding peer support initiatives, in which advice is given by experienced and trained peer counselors, is an effective way to promote and support breastfeeding, regardless of a woman's socioeconomic status. Several small studies have shown that breastfeeding peer support initiatives were effective for preterm infants and that this efficacy was increased by the co-intervention of lactation consultants.

The purpose of this study is to develop and to evaluate the effectiveness of a breastfeeding support program among mother-preterm infant dyads in Europe, by evaluating the impact of the intervention on 1) breastfeeding rates, 2) morbidity and mortality during the hospitalization, 3) children's cognitive development and behavior 4) mothers' mental health, 4) costs benefits.

The breastfeeding support program will include peer counselors under the supervision of lactation consultants. Breastfeeding counselors will be voluntary mothers who have had a positive breastfeeding experience with at least one preterm infant. After a training course, they will meet the future or new mothers by face-to-face and share their experiences at least once a week during hospitalization and provide phone support up to 1 month after discharge from hospital.

The study design will be a stepped wedge cluster trial conducted in 8 NICU in Europe (France, Switzerland and Belgium). Infants and mothers will be followed up from the time of hospitalization in the maternity and NICU up to 6 months after the discharge. The cost analysis will be performed in a subgroup of mother-preterm infant dyads that will be followed up at 24-months after their discharge

ELIGIBILITY:
Inclusion Criteria:

* any infant born <35 weeks' gestation,
* hospitalised in NICU before 24 hours old
* and younger than 168 hours (7 days) old.

Exclusion Criteria:

* infant with foetal malformation that is life-threatening
* infant with medical contraindication for breastfeeding
* parent(s)' non-consent to be involved in the study
* mother with prolonged medical contraindication for breastfeeding
* mother with psychiatric disorders making breastfeeding support impossible
* if no communication is possible with the mother
* if the level of communication with the mother does not allow breastfeeding support, with or without a third party

Max Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1774 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Breastfeeding continuation rates | at corrected postnatal age of 2 months
  Breastfeeding will be defined as the consumption of any mother's own milk. It will be classed as exclusive when all of the fed milk is the mother's own milk, or mixed when it will be completed by other milk and/or food.

SECONDARY OUTCOMES:
Rate of breastfeeding initiated | at 2 months of corrected age
Breastfeeding rate | at 2 months of corrected age
Breastfeeding rate | at the end of NICU stay
Breastfeeding rate | at 6 months of corrected age
Breastfeeding duration | at 6 months of corrected age
Neonatal severe complications | at 36 weeks of corrected age
  Morbidity outcomes will include intraventricular haemorrhage grade≥3, periventricular leucomalacia, sepsis (proven or clinical), persistent ductus arteriosus requiring treatment, necrotising enterocolitis grade≥2, and bronchopulmonary dysplasia (need of oxygen and/or ventilation support at 36 weeks of corrected age), retinopathy of prematurity grade>2.
Death rates | at 36 weeks of corrected age
  Morbidity outcomes will include intraventricular haemorrhage grade≥3, periventricular leucomalacia, sepsis (proven or clinical), persistent ductus arteriosus requiring treatment, necrotising enterocolitis grade≥2, and bronchopulmonary dysplasia (need of oxygen and/or ventilation support at 36 weeks of corrected age), retinopathy of prematurity grade>2.
Infant behaviours | at corrected postnatal age of 6 months
  Behavior will be assessed by the validated Infant Behavior questionnaire completed by mothers.
Mother-Infant bonding | at corrected postnatal age of 6 months
  Disabilities will include cerebral palsy, mental retardation assessed by the developmental quotient less than 85 on the Brunet- Lézine scale, and visual and hearing deficits. -Infant bonding assessed by the Mother-Infant Bonding Scale (MIBS)
Disability rate | at corrected postnatal age of 24 months
  Disabilities will include cerebral palsy, mental retardation assessed by the developmental quotient less than 85 on the Brunet- Lézine scale, and visual and hearing deficits.
Neurodevelopment rate by Brunet Lézine scale | at corrected postnatal age of 24 months
Anxiety by the Hospital Anxiety and Depression Scale (HADS) | at corrected postnatal age of 6 months
Depression by the Edinburgh Postnatal Depression Scale. | at corrected postnatal age of 6 months
Posttraumatic stress by the Post-traumatic stress disorder Checklist version DSM-5 (PCL-5) | at corrected postnatal age of 6 months
Parents stress by the Parenting Stress Index Fourth Edition Short Form (PSI-4 SF | at corrected postnatal age of 6 months
Costs effectiveness of breastfeeding | up to first two years of life
  Costs will include initial hospitalization, hospital readmissions, outpatient visits and tests.
cost consequence of breastfeeding | up to first two years of life
  Costs will include hospitalization rate and mortality between the two strategies.
Feasibility of the breastfeeding support program | 24 months
  To assess the feasibility of the intervention, we will depict : - the socio-demographic characteristics of breastfeeding counselors - and the number of contacts between mothers and breastfeeding counselors (frequency and duration) and the information
Acceptability of the breastfeeding support program | 24 months
  To assess the acceptability of the breastfeeding support program, we will collect :
  * the perception of breastfeeding support by mothers and their spouses, by staff members (lactation consultant, nurses) in each participating centers and by breastfeeding counselors.
  * the number of mothers who refuse to be managed by a breastfeeding counselors and their reasons,
  * the duration of each breastfeeding counselor intervention and the number of mothers who will stop the intervention before 1 month after the hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Laborie, MD, Principal Investigator — Hospices Civils de Lyon, Hôpital Femme Mère Enfant, Bron
Locations (8):
- CHC Clinique St-Vincent, Rocourt, Belgium
- France (6):
  - CHU site Félix Guyon, Saint-Denis, Réunion
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital Nord Ouest - Villefranche, Gleizé
  - CHU de Grenoble, Grenoble
  - CH Lyon Sud, Pierre-Bénite
  - Hôpital des Enfants, Toulouse
- CHU vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laborie S, Denis A, Horsch A, Occelli P, Margier J, Morisod Harari M, Claris O, Touzet S, Fischer Fumeaux CJ. Breastfeeding peer counselling for mothers of preterm neonates: protocol of a stepped-wedge cluster randomised controlled trial. BMJ Open. 2020 Jan 30;10(1):e032910. doi: 10.1136/bmjopen-2019-032910. PMID 32005780